CLINICAL TRIAL: NCT01781416
Title: Level of Concordance Between Patients Perception and Physicians Evaluation of Cardiovascular Risk
Acronym: PERCEPTION
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CFR-XXX-2012/1
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Risk
Keywords: cardiovascular risk; SCORE; cardiovascular primary prevention; risk factors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This is a national, non interventional, prospective study performed in the general practice setting.

The study has been designed :

* to assess the level of concordance between patients' cardiovascular risk perception and the cardiovascular risk evaluated by the physicians,
* and to evaluate the impact of patients' exposure to a medical information leaflet on patients' cardiovascular risk perception.

DETAILED DESCRIPTION:
LEVEL OF CONCORDANCE BETWEEN PATIENTS PERCEPTION AND PHYSICIANS EVALUATION OF CARDIOVASCULAR RISK

ELIGIBILITY:
Inclusion Criteria:

* Currently in primary prevention for a cardiovascular event (patient with no known history of acute cardiovascular or cerebrovascular event)
* Usually treated by the GP
* Having signed the information and consent form

Exclusion Criteria:

* Patient with a pathologic vascular ultrasound exam (atheromatous plaque or stenosis)
* Patient unable to read and complete the study documentation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adults aged 50 and over who :
  * are currently in primary prevention for a cardiovascular event,
  * are usually treated by the general practitioner,
  * and have a medical visit during the study period.
Sampling Method: Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk perceived by patients (before reading the Medical Information Leaflet) | Baseline
Cardiovascular risk assessed by physicians | Baseline

SECONDARY OUTCOMES:
Cardiovascular risks perceived by patients before and after reading the Medical Information Leaflet | Baseline
Actual cardiovascular risk calculated using SCORE | Baseline
Characteristics of patients whose self-evaluation of their CVR is concordant with their actual CVR | Baseline
Characteristics of patients whose self-evaluation of their CVR is discordant with their actual CVR | Baseline
Risk factors considered by patients in self-assessing their CVR | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Atul PATHAK, Professor, Study Chair — Service de Pharmacologie Clinique - Unite INSERM U 1048 - Faculte de Medecine - 37 Allees Jules Guesde -31073 Toulouse- FRANCE; Nicolas DANCHIN, Professor, Study Chair — Unite des Maladies Coronaires - Hopital Europeen Georges Pompidou - 20 Rue Leblanc - 75015 Paris - FRANCE
Locations (1):
- Research Site, Paris, France